CLINICAL TRIAL: NCT00185614
Title: Non-myeloablative Allogeneic Transplantation for the Treatment of Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wen-Kai Weng (Other)
Responsible Party: Sponsor-Investigator, Wen-Kai Weng, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13378; 75190 (Other: Stanford University Alternate IRB Approval No.); BMT109 (Other: OnCore)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Blood Cancer; Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma | interventions — Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Melphalan; Whole-Body Irradiation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Auto- then Allo-HCT (Experimental): Auto-HCT mobilization is cyclophosphamide 4 g/m2 + filgrastim 10 µg/kg/day for peripheral blood progenitor cell (PBPC) collection by apheresis. Transplant conditioning is high-dose melphalan 200 mg/m2, followed by PBPC infusion as melphalan rescue [ie, autologous hematopoietic cells transplant (Auto-HCT)]. Post-infusion support is filgrastim 5 µg/kg/day, starting 6 days after melphalan. Stable/responsive disease at 4 weeks continues to allogenic HCT (Allo-HCT) from sibling donor fully-matched for human leukocyte antigen (HLA). Allo-HCT conditioning is total body irradiation (TBI) 200 centigray (cGy) + cyclosporine (CSP) 6.25 mg/kg + mycophenolate mofetil (MMF) 15 mg/kg. Donor mobilization is filgrastim 16 µg/kg/day on day -4 to Day 0; apheresis collections on Day -1 & Day 0, to a target of > 5 x 10e6 CD34 cells/kg. Allo-HCT is infused to participant on Day 0, with premedication hydrocortisone 100 mg IV & diphenhydramine 50 mg IV. CSP tapering on Day 56 to Day 180, adjusted as needed.
  Interventions: Procedure: Autologous hematopoietic cell transplant (Auto-HCT); Procedure: Allogeneic hematopoietic cell transplant (Allo-HCT); Drug: Cyclophosphamide; Drug: Filgrastim; Drug: Melphalan; Radiation: Total body irradiation (TBI); Procedure: Cyclosporine (CSP); Drug: Mycophenolate Mofetil (MMF)

INTERVENTIONS:
Procedure: Autologous hematopoietic cell transplant (Auto-HCT) — The target cell dose is 2.6 x 10e6 CD34+ cells/kg
Procedure: Allogeneic hematopoietic cell transplant (Allo-HCT) — The target cell dose is 5 x 10e6 CD34 cells/kg
Drug: Cyclophosphamide — Cyclophosphamide administered intravenously (IV) at 4 mg /m² mobilize peripheral blood progenitor cells (PBPC) for autologous re-infusion
  Other Names: Cytoxan; Neosar
Drug: Filgrastim — * Filgrastim 10 µg/kg/day to mobilize peripheral blood progenitor cells (PBPC) for autologous re-infusion (Auto-HCT)
  * Filgrastim 5 µg/kg/day starting 6 days after melphalan (Day 4 after Auto-HCT)
  * Filgrastim 16 µg/kg/day to mobilize donor peripheral blood progenitor cells (PBPC) for allogeneic transplant (Allo-HCT)
  Other Names: Neupogen; Granulocyte-colony stimulating factor (G-CSF)
Drug: Melphalan — Melphalan 200 mg/m2 (high-dose) intravenously as conditioning for Auto-HCT
  Other Names: Melphalan hydrochloride; Melphalan HCl
Radiation: Total body irradiation (TBI) — 200 centigray (cGy) total body irradiation delivered on Day 0
Procedure: Cyclosporine (CSP) — Cyclosporine administered twice-daily by mouth at a dose of 6.25 mg/kg from Day -3 through Day 56
  Other Names: Cyclosporine A
Drug: Mycophenolate Mofetil (MMF) — Mycophenolate mofetil will begin at 15 mg/kg twice-daily by mouth from Day 0 to Day 27
  Other Names: CellCept

SUMMARY:
Mixed chimerism transplantation is an approach to allogeneic transplants that attempts to decrease regimen-related toxicity by using non-myeloablative preparatory regimens; establish mixed chimerism using low dose total body irradiation along with immunosuppression using cyclosporine and mycophenolate mofetil; suppress graft-vs-host and host-vs-graft reactions to allow a mixed chimeric state to be established, encourage tolerance and prevent graft-vs-host disease (GvHD) during the mixed chimerism period and use donor lymphocyte infusions to convert the patient to a full chimera while developing a graft-vs-tumor effect.

DETAILED DESCRIPTION:
Participants are mobilized with cyclophosphamide 4 g/m2 and filgrastim 10 µg/kg/day for peripheral blood progenitor cell (PBPC) collection by apheresis. Transplant conditioning is high-dose melphalan 200 mg/m2, followed by PBPC infusion as melphalan rescue [ie, autologous hematopoietic cells transplant (auto-HCT)]. Post-infusion support includes filgrastim 5 µg/kg/day, starting 6 days following melphalan. Participants with stable or responsive disease at 4 weeks eligible to continue on to the planned allogenic HCT (allo-HCT). For allo-HCT, a sibling donor that is fully matched for human leukocyte antigen (HLA-matched) is identified. Participants receive a single dose of total body irradiation (TBI) 200 centigray (cGy) as well as immunosuppression with cyclosporine (CSP) 6.25 mg/kg and mycophenolate mofetil (MMF) 15 mg/kg. The HLA-matched donor begins filgrastim injections 16 µg/kg/day on day -4 continuing to Day 0, with apheresis collections on Day -1 and Day 0, to a target of > 5 x 10e6 CD34 cells/kg. Allo-HCT is infused to participant on Day 0, with premedication hydrocortisone 100 mg IV and diphenhydramine 50 mg IV. CSP will be tapered beginning Day 56 with a goal of discontinuing CSP on Day 180, adjusted as needed.

ELIGIBILITY:
PATIENT INCLUSION CRITERIA

* Multiple myeloma, early Stage II-III or relapsed / progression after initial treatment of Stage I disease
* Patient has HLA-identical sibling donor
* Age ≤ 70 years
* No prior therapy which would preclude the use of low-dose total body irradiation
* Pathology review and diagnosis confirmation by Stanford University Medical Center
* Karnofsky performance status (KPS) > 70%
* DLCO ≥ 60% predicted
* ALT and AST < 2 x upper limit of normal (ULN)
* Total bilirubin < 2 mg/dL
* Serum creatinine < 2.0, or 24-hour creatinine clearance ≥ 60 mL/min
* HIV-negative
* Signed informed consent document

PATIENT EXCLUSION CRITERIA

* Smoldering multiple myeloma; monoclonal gammopathy of unknown significance; or primary amyloidosis
* Severe psychological or medical illness
* Prior allogeneic hematopoietic cell transplantation
* Pregnant or lactating

ALLOGENEIC DONOR INCLUSION CRITERIA

* Age ≥ 17
* HIV-seronegative
* Signed informed consent document

ALLOGENEIC DONOR EXCLUSION CRITERIA

* Serious medical or psychological illness
* Pregnant or lactating
* Prior malignancies within the last 5 years, except for non-melanoma skin cancers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2000-08; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kai Weng, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Autologous HCT (Auto-HCT)
Arm/Group | Auto- Then Allo-HCT
Started | 63
Completed | 63
Not Completed | 0
Period: Inter-treatment Period
Arm/Group | Auto- Then Allo-HCT
Started | 63 (Not all participants who received autologous transplant continued to receive allogeneic transplant.)
Completed | 59
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Relapse | 2
Not completed — Lack of allogenic donor | 1
Period: Allogenic HCT (Allo-HCT)
Arm/Group | Auto- Then Allo-HCT
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Auto- Then Allo-HCT
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 5
  White | 43
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: Event-free survival (EFS) as determined for all participants who received the initial Auto-HCT treatment. "Event" was defined as any of the following within 3 years of the participant's last infusion of Auto-HCT or Allo-HCT: relapse; death; or last follow-up if there is no data to document the participant remained alive at 3 years.
Time Frame: 3 years
Population: The outcome data are reported as the number of participants who do not experience an EFS event within 3 years from the date of the last transplant, for the "Auto-HCT only" population, the "Auto-HCT then Allo-HCT" population, and the overall study population (ie, "Auto-HCT only" plus +"Auto-HCT then Allo-HCT").
Measure: Count of Participants; unit: Participants
Arm/Group | Auto- Then Allo-HCT
Number analyzed (Participants) | 63
Participants
  Auto-HCT only: number analyzed (Participants) | 4
  Auto-HCT only | 0
  Auto-HCT then Allo-HCT: number analyzed (Participants) | 59
  Auto-HCT then Allo-HCT | 24
  All Participants | 24

2. Secondary Outcome: Relapse Rate
Description: Relapse rate as determined for all participants who received the initial Auto-HCT treatment. Relapse was protocol-specified as progressive disease, indicated by an increase as compared to pre-Auto-HCT baseline, of serum or urine monoclonal protein >25%; bone marrow plasmacytosis >25%; or bone lesions on skeletal survey (any increase).
Time Frame: 3 years
Population: The outcome data are reported as the number of participants who relapse per criteria within 3 years.
Measure: Number; unit: participants
Arm/Group | Auto- Then Allo-HCT
Number analyzed (Participants) | 63
participants
  Auto-HCT only: number analyzed (Participants) | 4
  Auto-HCT only | 2
  Auto-HCT then Allo-HCT: number analyzed (Participants) | 59
  Auto-HCT then Allo-HCT | 29
  All Participants | 31

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) as determined for all participants who received the initial Auto-HCT treatment, as assessed from the date of the last transplant.
Time Frame: 3 years
Population: The outcome data are reported as the number of participants who could be documented as remaining alive through 3 years from the date of the last transplant, for the "Auto-HCT only" population, the "Auto-HCT then Allo-HCT" population, and the overall study population (ie, "Auto-HCT only" plus +"Auto-HCT then Allo-HCT").
Measure: Number; unit: participants
Arm/Group | Auto- Then Allo-HCT
Number analyzed (Participants) | 63
participants
  Auto-HCT only: number analyzed (Participants) | 4
  Auto-HCT only | 1
  Auto-HCT then Allo-HCT: number analyzed (Participants) | 59
  Auto-HCT then Allo-HCT | 41
  All Participants | 42

4. Secondary Outcome: Acute Graft-vs-Host-Disease (aGvHD)
Description: Development of acute graft-vs-host-disease (aGvHD) within 6 months, for participants receiving Allo-HCT.
Time Frame: 6 months
Population: Graft versus host disease (aGvHD) only occurs in participants receiving Allo-HCT, as determined by investigator judgement (no protocol-specified criteria).
Measure: Count of Participants; unit: Participants
Arm/Group | Auto- Then Allo-HCT
Number analyzed (Participants) | 59
Participants | 7

5. Secondary Outcome: Chronic Graft-vs-Host-Disease (cGvHD)
Description: Development of chronic graft versus host disease (cGvHD) within 3 years, for participants receiving Allo-HCT. Reported as "Extensive cGvHD;" "cGvHD, Not Extensive;" or "No cGvHD," as determined by investigator judgement (no protocol-specified criteria).
Time Frame: 3 years
Population: Graft versus host disease (aGvHD) only occurs in participants receiving Allo-HCT.
Measure: Count of Participants; unit: Participants
Arm/Group | Auto- Then Allo-HCT
Number analyzed (Participants) | 59
Participants
  Extensive cGvHD | 30
  cGvHD, not Extensive | 8
  No cGvHD | 21

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- All Participants Receviing at Least Auto-HCT: Auto-HCT mobilization is cyclophosphamide 4 g/m2 + filgrastim 10 µg/kg/day for peripheral blood progenitor cell (PBPC) collection by apheresis. Transplant conditioning is high-dose melphalan 200 mg/m2, followed by PBPC infusion as melphalan rescue [ie, autologous hematopoietic cells transplant (Auto-HCT)]. Post-infusion support is filgrastim 5 µg/kg/day, starting 6 days after melphalan. Stable/responsive disease at 4 weeks continues to allogenic HCT (Allo-HCT) from sibling donor fully-matched for human leukocyte antigen (HLA). Allo-HCT conditioning is total body irradiation (TBI) 200 centigray (cGy) + cyclosporine (CSP) 6.25 mg/kg + mycophenolate mofetil (MMF) 15 mg/kg. Donor mobilization is filgrastim 16 µg/kg/day on day -4 to Day 0; apheresis collections on Day -1 & Day 0, to a target of > 5 x 10e6 CD34 cells/kg. Allo-HCT is infused to participant on Day 0, with premedication hydrocortisone 100 mg IV & diphenhydramine 50 mg IV. CSP tapering on Day 56 to Day 180, adjusted as needed.
Arm/Group | All Participants Receviing at Least Auto-HCT
All-Cause Mortality (participants affected / at risk) | 21/63
Serious Adverse Events (participants affected / at risk) | 63/63
Other Adverse Events (participants affected / at risk) | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Receviing at Least Auto-HCT (N=63)
Lung Aspergillosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Heart Failure (Cardiac disorders) | 1 (1)
Cardiopulmonary Failure (Cardiac disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Aseptic Encephalitis (Psychiatric disorders) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2)
Cytomegalovirus (Immune system disorders) | 2 (2)
Coagulase-negative staphylococci (Blood and lymphatic system disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Disseminated varicella zoster (Skin and subcutaneous tissue disorders) | 4 (4)
Erosive esophagitis (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 31 (31)
Fever (Infections and infestations) | 3 (3)
Fungemia (Blood and lymphatic system disorders) | 1 (1)
Gram-negative bacillary bacteremia (Blood and lymphatic system disorders) | 6 (6)
Herpetic stomatitis (Nervous system disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Klebsiella bacteremia (Infections and infestations) | 1 (1)
Lung Aspergillosis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Mucositis (Gastrointestinal disorders) | 8 (8)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Platelet count decrease (Blood and lymphatic system disorders) | 3 (4)
Pneumonia (Infections and infestations) | 2 (2)
Pseudomonas bacteremia (Blood and lymphatic system disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Rhabdomyositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Parietal Encephalocele (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory syncytial virus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Superior Vena Cava Syndrome (Cardiac disorders) | 1 (1)
Viral Pneumonitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Receviing at Least Auto-HCT (N=63)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Ascites (Renal and urinary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cytomegalovirus (Immune system disorders) | 5 (6)
Coagulase-negative staphylococci (Blood and lymphatic system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehyration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Disseminated varicella zoster (Skin and subcutaneous tissue disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 5 (5)
Fever (Infections and infestations) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Herpes Zoster (Nervous system disorders) | 1 (1)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 6 (6)
Mucositis (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 16 (17)
Parainfluenza pneumonitis (Infections and infestations) | 1 (1)
Platelet count decrease (Blood and lymphatic system disorders) | 14 (15)
Renal Failure (Renal and urinary disorders) | 15 (16)
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Steroid Myopathy (Gastrointestinal disorders) | 1 (1)
Transaminitis (Blood and lymphatic system disorders) | 1 (1)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 2 (2)
Viral bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Viral Pneumonitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No